CLINICAL TRIAL: NCT04118127
Title: A Multi-center, Open-label Clinical Pharmacology Trial to Investigate the Pharmacokinetics, Tolerability, and Safety of Brexpiprazole Once-weekly (QW) Formulation Administered as Single and Multiple Oral Doses in Patients With Schizophrenia
Brief Title: A Clinical Pharmacology Trial of Brexpiprazole Once-weekly (QW) Formulation Administered as Single and Multiple Oral Doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-102-00150
Record Dates: First submitted 2019-10-04; First posted 2019-10-08 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia,brexpiprazole,open-label,linical pharmacology
MeSH Terms: conditions — Schizophrenia | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2mg conventional tablet, once-weekly tablets (Experimental)
  Interventions: Drug: 2mg conventional tablet, once-weekly tablets

INTERVENTIONS:
Drug: 2mg conventional tablet, once-weekly tablets — In each cohort, subjects will receive a brexpiprazole 2 mg conventional tablet on Day 1of Period 1, the QW formulation on Day 1 of Period 2 and 3, as single and multiple dose in a fasted state.

SUMMARY:
To evaluate the pharmacokinetics (PK), tolerability, and safety of brexpiprazole QW formulation administered as single and multiple doses in patients with schizophrenia.

DETAILED DESCRIPTION:
A multi-center, open-label clinical pharmacology trial to investigate the PK, tolerability, and safety of brexpiprazole QW formulation administered as single and multiple doses.

The trial comprises the single-dose period (Cohort 1) and the multiple-dose period (Cohort 2). The dose used in the multiple-dose period (Cohort 2) will be determined based on plasma drug concentrations obtained in the single-dose period (Cohort 1).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of schizophrenia based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
2. Patients capable of staying at the trial site from the day before investigational medicinal product (IMP) administration to the 8th day following IMP administration in both Period 1 and Period 2
3. Patients with a body mass index [BMI = body weight (kg)/height (m)2] of 18.5 or higher and lower than 35.0 at screening
4. Persons who provide written informed consent before commencement of any trial-related procedures and whom the investigator or subinvestigator judges to be capable of following all the conditions of this trial
5. Patients who, in the judgement of the investigator or subinvestigator, have stable psychotic symptoms maintained by administration of an antipsychotic (other than clozapine) within the dosing range indicated separately, before commencement of investigational medicinal product (IMP) administration"

Exclusion Criteria:

1. Patients with a diagnosis of a concurrent mental disorder besides schizophrenia (schizoaffective disorder, major depressive disorder, bipolar I disorder, bipolar II disorder, general anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, dementia or mild neurocognitive disorder, personality disorder, etc) based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) (However, this exclusion does not apply to caffeine- or tobacco-related disorders)
2. Patients who fail to meet the specified requisite washout periods for the prohibited concomitant drugs and foods before commencement of IMP administration, or patients who are anticipated to take any of these drugs or foods during the study period
3. Patients who have previously undergone gastrointestinal surgery that could affect pharmacokinetic evaluations
4. Patients who are using clozapine at the time of informed consent
5. Patients who have received electro-convulsive therapy within 60 days before commencement of IMP administration
6. Patients with clinically problematic disorders of the nervous system, liver, kidneys, metabolic system, blood, immune system, cardiovascular system, lungs, or digestive system (However, such patients may be included if the condition is mild or well-controlled and is considered to not affect safety or pharmacokinetic evaluations.)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Sankeikai Nishigahara Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total number of subjects who participated in Cohort 1 and Cohort 2 was 73.
Groups:
- Cohort 2: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1. Subjects washed out brexpiprazole for 20 days until Period 2(Cohort 2). Subjects received a brexpiprazole QW formulation at 24 mg on Day 1. Subjects repeated administration of the QW formulation at 48 mg on Days 8, 15, 22, and 29.
- Cohort 1: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1. Subjects washed out brexpiprazole for 20 days until Cohort 1 Period 2. Subjects received a brexpiprazole QW formulation at 24 mg on Day 1. Subjects washed out brexpiprazole for 27 days until Cohort 1 Period 3. Subjects received a brexpiprazole QW formulation at 48 mg on Day 1
Period: Overall Study
Arm/Group | Cohort 2 | Cohort 1
Started | 35 | 38
Completed | 32 | 22
Not Completed | 3 | 16
Not completed — Trial terminated by sponsor | 0 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: The total number of subjects who participated in Cohort 1 and Cohort 2 was 73. The total age average was calculated from 73 subjects in period 1 of Cohort 1 and Cohort 2.
Groups:
- Cohort 1 Period 1: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1. Subjects washed out brexpiprazole for 20 days until Cohort 1 Period 2.
- Cohort 2 Period 1: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1. Subjects washed out brexpiprazole for 20 days until Period 2(Cohort 2).
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Period 1 | Cohort 2 Period 1 | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (9.7) | 47.1 (10.6) | 46.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 24 | 19 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 38 | 35 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of OPC-34712 Following Single Oral Administration of 24 mg and 48 mg QW Formulation or 2 mg Conventional Tablet in Cohrt1
Description: To evaluate Cmax of OPC-34712 following single oral administration of the QW formulation (24 mg and 48 mg) and 2 mg conventional tablet .
Time Frame: prepose, 2,4, 6, 8, 12, 24, 48, 72, 120, 168, 240, 312 hours postdose
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Conventional Tablet 2mg: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1.
- QW Formuration 24mg: Subjects received a brexpiprazole QW formulation at 24 mg on Day 1.
- QW Formuration 48mg: Subjects received a brexpiprazole QW formulation at 48 mg on Day 1
Arm/Group | Conventional Tablet 2mg | QW Formuration 24mg | QW Formuration 48mg
Number analyzed (Participants) | 33 | 33 | 22
ng/mL | 25.37 (10.46) | 98.62 (46.76) | 222.3 (114.3)

2. Primary Outcome: Time to Maximum (Peak) Plasma Concentration (Tmax) of OPC-34712 Following Single Oral Administration of 24 mg and 48 mg QW Formulation or 2 mg Conventional Tablet in Cohrt1
Description: To evaluate Tmax of OPC-34712 following single oral administration of the QW formulation (24 mg and 48 mg) and 2 mg conventional tablet .
Time Frame: prepose, 2,4, 6, 8, 12, 24, 48, 72, 120, 168, 240, 312 hours postdose
Measure: Median (Full Range); unit: hour
Arm/Group | Conventional Tablet 2mg | QW Formuration 24mg | QW Formuration 48mg
Number analyzed (Participants) | 33 | 33 | 22
hour | 4.00 [1.75 to 24.37] | 25.37 [8.75 to 49.50] | 25.00 [8.60 to 46.42]

3. Primary Outcome: Cmax of OPC-34712 Following Multiple Oral Administrations of 48 mg QW Formulation in Cohort 2 Period 2
Description: To evaluate Tmax of OPC-34712 following multiple oral administration of the QW formulation 48 mg.
Time Frame: prepose, 3, 9, 24, 36, 48, 72, 120, 168, 240, 312 hours postdose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | QW Formuration 48mg
Number analyzed (Participants) | 32
ng/mL | 225.0 (147.7)

4. Primary Outcome: Tmax of OPC-34712 Following Multiple Oral Administrations of 48 mg QW Formulation in Cohort 2 Period 2
Description: To evaluate Tmax of OPC-34712 following multiple oral administration of the QW formulation 48 mg.
Time Frame: prepose, 3, 9, 24, 36, 48, 72, 120, 168, 240, 312 hours postdose
Measure: Median (Full Range); unit: hour
Arm/Group | QW Formuration 48mg
Number analyzed (Participants) | 32
hour | 24.61 [8.50 to 49.25]

ADVERSE EVENTS:
Time Frame: From the start of IMP administration throughout follow-up period Cohort 1: up to 93 days (Period 1: up to 28 days, Period 2: up to 35 days, Period 3: up to 30 days) Cohort 2: up to 88 days (Period 1: up to 28 days, Period 2: up to 60 days)
Description: Adverse events (AEs) in each participant were monitored in each period of Cohort 1 and 2, with the maximum duration as indicated above, from after the IMP administration in each period until before the IMP administration in the next period (for Cohort 1 period 1-2 and Cohort 2 period 1) or the end of study (for Cohort 1 period 3 and Cohort 2 period 2). AEs were assessed separately in Cohort 1 (period 1-3) and Cohort 2 (period 1-2).
Groups:
- Cohort 1 Period 2: Subjects received a brexpiprazole QW formulation at 24 mg on Day 1. Subjects washed out brexpiprazole for 27 days until Period 3(Cohort 1).
- Cohort 1 Period 3: Subjects received a brexpiprazole QW formulation at 48 mg on Day 1
- Cohort 2 Period 2: Subjects received a brexpiprazole QW formulation at 24 mg on Day 1. Subjects repeated administration of the QW formulation at 48 mg on Days 8, 15, 22, and 29.
- Cohort 2 Period 1: Subjects received a brexpiprazole 2 mg conventional tablet on Day 1. Subjects washed out brexpiprazole for 20 days until Cohort 2 Period 2.
Arm/Group | Cohort 1 Period 2 | Cohort 1 Period 3 | Cohort 2 Period 2 | Cohort 1 Period 1 | Cohort 2 Period 1
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/23 | 0/34 | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/23 | 0/34 | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 21/34 | 11/23 | 20/34 | 16/38 | 16/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Period 2 (N=34) | Cohort 1 Period 3 (N=23) | Cohort 2 Period 2 (N=34) | Cohort 1 Period 1 (N=38) | Cohort 2 Period 1 (N=35)
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Period 2 (N=34) | Cohort 1 Period 3 (N=23) | Cohort 2 Period 2 (N=34) | Cohort 1 Period 1 (N=38) | Cohort 2 Period 1 (N=35)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 1 | 0 | 1 | 0 | 0
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 1
Thirst (General disorders) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected Dermal Cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 2 | 2 | 2
Oral Herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 3 | 0 | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 1 | 0 | 0
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 2 | 0 | 0
Blood Glucose Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Insulin Increased (Investigations) | 1 | 1 | 0 | 0 | 2
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Pressure Decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Pressure Systolic Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Prolactin Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Urinary Occult Blood Positive (Investigations) | 1 | 1 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight Increased (Investigations) | 0 | 0 | 1 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle Rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 2 | 3 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dystonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Extrapyramidal Disorder (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 4 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Mental Impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Restless Legs Syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 4 | 2 | 1
Taste Disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0
Hallucination (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Menstrual Disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Faeces Hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Injection Site Pruritu (General disorders) | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Triglycerides Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Uric Acid Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Vagus Nerve Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Scrotal Dermatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT04118127/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/27/NCT04118127/SAP_001.pdf